CLINICAL TRIAL: NCT05370677
Title: The Prevelence of IVS 1-6 (T-C) [HBB:c.92 +6 T-C] Gene Mutation in Suspected Cases of β Thalassemia in Assiut University Hospitals
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Fatma Elzahraa Mohamed Abd Elrady Farghly, resident doctor, Assiut University
Other Study IDs: thalassemia mutation
Record Dates: First submitted 2022-05-07; First posted 2022-05-11 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Beta-Thalassemia
MeSH Terms: conditions — beta-Thalassemia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: ARMS — amplification refractory mutation system

SUMMARY:
1. - To design an amplification-refractory mutation system (ARMS) for the DNA diagnosis of the IVS I-6 (T>C) mutation.
2. - To detect the prevelence of the mutation among Assiut University Hospital patients.
3. - Phenotype/genotype correlation of the mutation.

DETAILED DESCRIPTION:
• The β-thalassaemias result from 300 gene mutations ( https://globin.bx.psu.edu ).

All of the mutations are regionally specific and the spectrum of mutations has now been determined for most at-risk populations(Old JM, 2007).

* The strategy for identifying β-thalassaemia mutations is usually based on the knowledge of the common and rare mutations in the ethnic group of the individual being screened.(Old JM, 2007) .
* In Mediterranean it represnts 8-15%
* In Africa it represnts 3.5%
* In Egyptians it represnts 13.6% ( https://globin.bx.psu.edu ).
* The β globin gene mutation IVS I-6(T>C) is the First most common β globin gene mutation among Egyptians
* (36.3%) according to ( Somaia El-Gawhary et al 2007 )
* (27.66%) ( Ammar D. Elmezayen et al 2015 )
* and the second most common mutation
* (40%) according to ( El-shanshory M et al 2014)
* (21.25%) ( Elhalfawy et al 2017) The molecular characterization of the globin gene mutation is necessary for definite diagnosis, genetic counseling, and to offer prenatal diagnosis. The amplification-refractory mutation system (ARMS) is a simple method for detecting any mutation involving single base changes or small deletions.
* the DNA is analysed after amplification by PCR for Detection of point mutation IVS I-6(T>C) by Using primer pairs that only amplify individual alleles [ARMS] .

ELIGIBILITY:
Inclusion Criteria:

* : β thalassemia (suspected & clinically diagnosed cases).

Exclusion Criteria:

* : Iron deficiency anaemia, anaemia of chronic disease, types of haemolytic anaemias other than thalassemia, other types of thalassemia and Hb variants

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: around 141 (suspected & clinically diagnosed cases).
Sampling Method: Non-Probability Sample
Enrollment: 141 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
using ARMS to detect the mutation | 2 years
  * To introduce the ARMS PCR as a cheap and simple DNA diagnostic tool for any point mutation.
  * Initiating the department database of haemoglobinopathesis by regisptering data.

SECONDARY OUTCOMES:
teaching purpose | 2 years
  teaching purpose

REFERENCES:
- [Background] Origa R. beta-Thalassemia. Genet Med. 2017 Jun;19(6):609-619. doi: 10.1038/gim.2016.173. Epub 2016 Nov 3. PMID 27811859
- [Background] Galanello R, Origa R. Beta-thalassemia. Orphanet J Rare Dis. 2010 May 21;5:11. doi: 10.1186/1750-1172-5-11. PMID 20492708
- [Background] Kumar R, Sagar C, Sharma D, Kishor P. beta-globin genes: mutation hot-spots in the global thalassemia belt. Hemoglobin. 2015;39(1):1-8. doi: 10.3109/03630269.2014.985831. Epub 2014 Dec 19. PMID 25523871
- [Background] Hashmi G, Qidwai A, Fernandez K, Seul M. Enabling routine beta-thalassemia Prevention and Patient Management by scalable, combined Thalassemia and Hemochromatosis Mutation Analysis. BMC Med Genet. 2020 May 15;21(1):108. doi: 10.1186/s12881-020-01017-x. PMID 32414341